CLINICAL TRIAL: NCT02535533
Title: A Therapeutic Trial for Safety and Preliminary Efficacy of the Combination of Axitinib and Seleniomethionine (SLM) for Adult Patients With Advanced Metastatic Clear Cell Renal Cell Carcinoma (CCRCC)
Brief Title: SLM + Axitinib for Clear Cell RCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mohammed Milhem (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Mohammed Milhem, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201507716
Record Dates: First submitted 2015-08-17; First posted 2015-08-28 (Estimated); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Advanced Metastatic Clear Cell Renal Cell Carcinoma (CCRCC)
Keywords: Kidney cancer; Selenium (Se)
MeSH Terms: conditions — Kidney Neoplasms | interventions — Selenomethionine; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Treatment (Experimental): During the Dose-Escalation Part 1, patients will receive SLM twice daily for 14 days followed by SLM once daily in combination with axitinib 5 mg twice daily with titration according to package insert. Treatment will continue until disease progression or unacceptable toxicity.
  During the Expansion Part 2, patients will be treated at the maximum tolerated dose (MTD) of SLM determined as 4000 mcg SLM. SLM will be given orally twice daily for 14 days followed by SLM once daily in combination with axitinib 5 mg twice daily with titration according to package insert. Treatment will continue until disease progression or unacceptable toxicity.
  During the Pilot Phase, dosing will begin at dose level 3 (4000, 5000, or 6000 mcg SLM calculated based on patients' BSA). SLM will be given orally twice daily for 14 days. Each cohort will enroll 2 evaluable patients.
  Interventions: Drug: Selenomethionine (SLM); Drug: Axitinib

INTERVENTIONS:
Drug: Selenomethionine (SLM) — SLM administrated orally twice daily for 14 days followed by SLM once daily in combination with Axitinib 5 mg twice daily with titration according to package insert
Drug: Axitinib — Following SLM administrated orally twice daily for 14 days, SLM once daily in combination with Axitinib 5 mg twice daily with titration according to package insert
Drug: Selenomethionine (SLM) — Maximum tolerated dose (MTD) of SLM determined in the Escalation Part 1 (4000 mcg SLM) given orally twice daily for 14 days, followed by SLM once daily in combination with axitinib 5 mg twice daily with titration according to package insert
Drug: Axitinib — Following maximum tolerated dose (MTD) of SLM determined in the Escalation Part 1 (4000 mcg SLM) given orally twice daily for 14 days, SLM once daily in combination with axitinib 5 mg twice daily with titration according to package insert
Drug: Selenomethionine (SLM) — Pilot Phase - Dosing will begin at dose level 3 (4000, 5000 or 6000 mcg SLM calculated based on patients' BSA). SLM will be given orally twice daily for 14 days

SUMMARY:
This phase I trial studies the side effects and best dose of L-selenomethionine when given together with axitinib in treating patients with clear cell renal cell carcinoma that has spread from the primary site (place where it started) to other places in the body and usually cannot be cured or controlled with treatment (advanced metastatic). L-selenomethionine may stop the growth of tumor cells by blocking the growth of new blood vessels necessary for tumor growth. Axitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving L-selenomethionine together with axitinib may be a better treatment for advanced metastatic clear cell renal cell carcinoma.

DETAILED DESCRIPTION:
This is a Phase I trial for safety and preliminary efficacy of the combination of axitinib and SLM for adult patients with advanced metastatic CCRCC. This will be a two part study consisting of a dose escalation and expansion study.

Dose-Escalation Part 1 (6-12 patients): SLM will be given twice daily for 14 days followed by once daily dosing in combination with axitinib 5 mg twice daily with titration according to package insert in patients with advanced renal cell carcinoma. Treatment will continue until disease progression or unacceptable toxicity. The MTD was determined to be 4000 mcg SLM.

Expansion Part 2: In this phase (approximately 19 patients), will be treated at the maximum tolerated dose (MTD) of SLM determined in the Escalation Part 1. It will be given orally twice daily for 14 days, followed by once daily dosing in combination with axitinib 5 mg twice daily with titration according to package insert in patients with advanced renal cell carcinoma. Treatment will continue until disease progression or unacceptable toxicity.

A pilot group of 10 subjects will have SLM dose calculated based on patients' BSA to characterize the dose-concentration relationship and estimate the effective administered dose of selenium necessary to achieve the target blood concentration range informed by preclinical data.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following criteria to be enrolled in this study:

* Histologically and radiologically confirmed advanced metastatic CCRCC in patients who have had at least one prior systemic therapy, which can include axitinib for the dose escalation part. In the expansion and pilot phases, patients with prior axitinib are allowed, as long as the last dose of axitinib was longer than 6 months ago.
* Written and voluntary informed consent.
* At least one Response Evaluation Criteria In Solid Tumors (RECIST)-defined target lesion. *Patient must have documented disease progression.
* Renal function (creatinine level within normal institutional limit, or creatinine clearance >15 mL/min/1.73 m2 for patients with creatinine levels above institutional normal, calculated using the Cockcroft-Gault formula).
* Liver function (AST/ALT <2.5 X institutional upper limit of normal OR < 5 x institutional upper limit of normal in cases of liver metastases; Total bilirubin ≤ 1.5 times ULN.)
* Adequate hematological lab values including;

  * Absolute Neutrophil Count (ANC) ≥ 1.0 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hemoglobin ≥ 7.0 g/dL
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 (fully active, able to carry on all pre-disease performance without restriction), 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, such as light housework or office work) or 2 (Ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours).
* Age of at least 18 years.
* Life expectancy of 12 weeks and more.
* 2 weeks or more since end of previous systemic treatment (4 weeks or more for bevacizumab plus interferon-alfa). 3 days wash out for palliative radiation.
* Must have a safely accessible biopsy per treating physician and the provider performing that biopsy. Patient must agree to have this biopsy done as outlined in the calendar. If patient does not have safely accessible biopsy, the patient may still be enrolled per investigator discretion.

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

* Patients with prior malignancies of the same or different tumor type in the last 5 years and patients with concurrent malignancies of the same or different tumor type UNLESS the natural history of the disease or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational drug.
* Symptomatic untreated metastases in the central nervous system.
* Subject that is pregnant or lactating.
* Pre-existing uncontrolled hypertension defined as > 150/90 mm Hg with medication.
* Present use or anticipated need for cytochrome P450 (CYP) 3A4-inhibiting, CYP3A4-inducing drugs (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, and voriconazole, rifampin, phenytoin, carbamazepine, rifabutin, rifapentin, phenobarbital, and St. John's wort, bosentan, efavirenz, etravirine, modafinil, and nafcillin).Myocardial infarction, uncontrolled angina, congestive heart failure, or cerebrovascular accident within previous 6 months. Subjects with history of deep vein thrombosis or pulmonary embolism, at provider discretion.
* Major surgery within 4 weeks of starting study treatment.
* Known HIV or acquired immunodeficiency syndrome-related disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) per CTCAE 4.03 | After 2 cycles (28 days)
  The AEs will be summarized and classified by body system and by treatment group. The type, incidence, severity, and causality of each AE, the duration of the event, and any required treatment interventions will be tabulated.
Pilot Phase - Determine dose-concentration relationship and estimate the effective dose of SLM (informed by preclinical data) using the continual reassessment method (CRM). | 14 days
  Dose escalation for this pilot study will be conducted using a CRM in which the probability of exceeding a blood selenium concentration of 45 µM on Day 14 is being modeled. Prior probabilities of exceeding a blood selenium concentration of 45 µM on Day 14 were estimated based on preclinical and preliminary data from the initial trial. A one parameter logistic model with intercept set at 3 and an initial value of 1 for the slope will be used to estimate the dose-concentration relationship through sequential recursive Bayesian assessment. The target probability of exceeding 45 µM is ≤20%.

SECONDARY OUTCOMES:
Tumor Response rate as assessed by RECIST v.1.1 | After 2 cycles (28 days)
Progression free survival (PFS) | 14 months
Overall survival (OS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milhem, MBBS, Principal Investigator — University of Iowa Hospitals & Clinics
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT02535533/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT02535533/ICF_001.pdf